CLINICAL TRIAL: NCT05313126
Title: Immuno-epidemiological and Socio-behavioral Evaluation of Release of Sterile Male Aedes Albopictus Mosquitoes on Human-vector Contacts
Acronym: EXPOCAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-A03558-31
Record Dates: First submitted 2022-01-05; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Mosquito Bite

STUDY DESIGN:
Intervention Model Description: A Cluster-Non Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sterile male Aedes albopictus-exposed (Experimental): Sterile male Aedes albopictus are released in the area.
  Interventions: Other: sterile insect technique (TIS)
- control (No Intervention): Sterile male Aedes albopictus are not released in the area.

INTERVENTIONS:
Other: sterile insect technique (TIS) — Sterile male Aedes albopictus mosquitos are released in the area/neighborhood
  Arms: sterile male Aedes albopictus-exposed

SUMMARY:
This trial is based on 2 complementary components, named ExpAlbo Biomarker and CAPAlbo Questionnaire

1. ExpAlbo Biomarker (Exposure to the Aedes albopictus mosquito): This component concerns the epidemiological evaluation of the effectiveness of the release of sterile male mosquitoes on the level of exposure of individuals to the bites of the tiger mosquito through the use of a new immunological biomarker of the human-vector contact, developed over the past 20 years by the IRD-MIVEGEC team. Indeed, when a person is bitten by a mosquito, he or she develops a defence reaction, called an immune reaction, against the mosquito's saliva. The main objective of this study is to measure this immune response, and more specifically the antibody response specifically directed against compounds (peptide = small fragment of a protein) in mosquito saliva, and to determine whether this anti-saliva antibody response, and therefore exposure to mosquito bites, decreases when the mosquito control strategy is applied.
2. CAPAlbo Questionnaire: This component is concerned with assessing the impact of sterile male mosquito releases on perceptions and practices related to exposure to Aedes albopictus based on population-based questionnaire surveys. The main objective of these surveys is to determine whether changes in objective exposure to Aedes albopictus mosquitoes are associated with changes in the perception of the nuisance and in the lifestyle habits of respondents, particularly those related to the prevention of mosquito bites (such as the use of repellents or mosquito nets).

ELIGIBILITY:
Inclusion Criteria:

* To inhabit on a regular basis in the intervention/control area
* To speak French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Immunological indicators | 6 months
  Biomarker based on the measurement of human IgG antibody levels specific to one peptide of Aedes saliva (i.e. Nterm-24kDa salivary peptide)
Immunological indicators | 12 months
  Biomarker based on the measurement of human IgG antibody levels specific to one peptide of Aedes saliva (i.e. Nterm-24kDa salivary peptide)
Exposure to Aedes mosquito | 6 months
  self-perceived exposure to mosquito will be assessed by questionnaire
Exposure to Aedes mosquito | 12 months
  self-perceived exposure to mosquito will be assessed by questionnaire

SECONDARY OUTCOMES:
Protective behavior | 6 months
  a composite indicator derived from a questionnaire will rate the protective behavior of the participants to avoid mosquito bites
Protective behavior | 12 months
  a composite indicator derived from a questionnaire will rate the protective behavior of the participants to avoid mosquito bites

CONTACTS AND LOCATIONS:
Locations (1):
- population générale (quartier Duparc (Sainte Marie) et Quartier Bois rouge), La Réunion, France

IPD SHARING:
Plan to Share IPD: Undecided